CLINICAL TRIAL: NCT02162277
Title: Phase 1 Study of Osteoporotic Diagnosis Using Osteoporotic Diagnostic Kits
Brief Title: Therapeutic Strategy in Postmenopausal Women Using Osteoporotic Diagnostic Kits
Status: Completed | Type: Observational
Sponsor: Shinshu University (Other)
Responsible Party: Principal Investigator, Yukio Nakamura, Assistant professor, Shinshu University
Other Study IDs: Showa-Hitachi2014; Osteoporotic diagnostic kit (Other: Showa Inan General Hospital)
Record Dates: First submitted 2014-06-09; First posted 2014-06-12 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Osteoporosis
Keywords: To decrease; number; osteoporotic; patients in; Kami-Ina area; Nagano prefecture
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Osteoporosis diagnostic kit
  Interventions: Device: diagnostic osteoporotic kit ( including 7 genes and 4 life styles)

INTERVENTIONS:
Device: diagnostic osteoporotic kit ( including 7 genes and 4 life styles) — Most osteoporotic patients want to know what kinds of life styles they should take care of. The device will help it.

SUMMARY:
The frequency of osteoporosis in Japan is increasing. Also, the frequency of osteoporosis-based fractures in postmenopausal women is increasing. Therefore, it is urgently required to improve osteoporosis. Life expectancy in Nagano prefecture is the longest in Japan, however, healthy life expectancy in Nagano is not very long in Japan. There are several problems in this issue from the medical site and the patient site. The aim of this study is, from the patient site, to increase the motivation of postmenopausal women for osteoporosis using osteoporotic diagnostic kit.

ELIGIBILITY:
Inclusion Criteria:

* Women, mainly postmenopausal women

Exclusion Criteria:

* Men

Ages: 20 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who are over 20 years old
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2013-01 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with osteoporosis in Kami-Ina area of Nagano prefecture | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Yukio Nakamura, Matsumoto, Nagano, Japan